CLINICAL TRIAL: NCT00229697
Title: A Phase II Randomised, Double-Blind, Stratified, Multi-Centre Trial Comparing the Nolvadex 20 Mg And Placebo Combination To The Nolvadex 20 Mg and ZD1839 (IRESSA™) 250 MG Combination In Patients With Metastatic Breast Cancer And Estrogen Receptor (ER) and/or Progesterone (PR) Positive Tumours
Brief Title: Phase II Metastatic ER+/PgR+ Nolvadex +/- Iressa Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1839IL/0225; D7917C00225; NCT00069290 (obsolete NCT alias)
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): ZD1839 + Nolvadex
  Interventions: Drug: Gefitinib; Drug: Tamoxifen
- 2 (Other): Nolvadex + placebo
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Gefitinib
  Other Names: Iressa
  Arms: 1
Drug: Tamoxifen
  Other Names: Nolvadex

SUMMARY:
This study is being carried out to see if ZD1839 is effective in treating metastatic breast cancer in combination with Nolvadex, and if so, how it compares with Nolvadex alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic adenocarcinoma of the breast (seeTNM staging Appendix I) that is ER and/or PR positive as determined in local laboratories at each investigator site (central verification of ER status will be performed after the patient starts treatment
* A tissue block from either the metastatic or primary tumor site is required.
* WHO performance status (PS) 0-2
* Patients must not be pregnant or breast-feeding. A negative pregnancy test is required within 7 days prior to randomization if pre- or peri-menopausal. Postmenopausal patients are defined as:
* natural menopause with last menses > 1 year ago,
* radiation induced oophorectomy with last menses > 1 year ago,
* chemotherapy induced menopause with 1 year interval since last menses, or
* serum FSH and LH and plasma estradiol levels in the postmenopausal range for the institution.
* bilateral oophorectomy

Exclusion Criteria:

* Patients cannot be on hormone replacement therapy or received prior chemotherapy for metastatic disease.
* Patients previously treated with a Tyrosine Kinase inhibitor or have evidence of an active interstitial lung disease are not eligible.
* Treatment with LH-RH analog.
* Laboratory values as follow Bilirubin >1.5 times upper limit of normal ULN, alanine amino transferase (ALT) or aspartate amino transferase (AST) >2.5 times the ULN if no demonstrable liver metastases, or >5 times the ULN in the presence of liver metastases
* Bone marrow function: WBC <1500 mm3

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2003-10; Primary Completion 2006-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Strata 1: To compare the time to progression between 2 treatment arms (ZD1839/Nolvadex vs placebo/Nolvadex) | Time to progression (progressive disease or death; equivalent to progression-free survival)
Strata 2: To compare the clinical benefit rate between 2 treatment arms (ZD1839/Nolvadex vs placebo/Nolvadex) | Overall clinical benefit rate: Complete Response, Partial Response or Stable Disease > 24weeks after each combination

SECONDARY OUTCOMES:
To compare the clinical benefit rate between 2 treatment arms (ZD1839/Nolvadex vs placebo/Nolvadex) in Strata 1 and overall | Overall clinical benefit rate: Complete Response, Partial Response or Stable Disease >24 weeks after each combination. Objective tumour resp defined according to RECIST criteria
To compare time to progression between 2 treatment arms (ZD1839/Nolvadex vs placebo/Nolvadex) in Strata 2 and overall | Time to progression (progressive disease or death)
To compare the objective response rate between ZD1839/Nolvadex and placebo/Nolvadex in each strata and overall | Objective tumour response (OR) defined according to RECIST criteria
To estimate duration of response for the ZD1839/Nolvadex and placebo/Nolvadex treatments in each strata and overall | Duration of response (CR and PR)
To compare overall survival between the ZD1839/Nolvadex and placebo/Nolvadex in each strata | Overall survival
To assess whether patients with high tumour levels of HER-2 and/or AIB1 demonstrate de novo resistance to Nolvadex therapy or have shorter TTP or response duration when compared with Nolvadex/ZD1839 treatment | Time to progression (progressive disease or death), duration of response (CR and PR)
To compare the objective response rate between the ZD1839/Nolvadex and placebo/Nolvadex treatment arms in the subset of all patients with ER+ tumours staining 2+/3+ for Her2neu by IHC | Objective tumour response (OR) defined according to RECIST criteria
To compare the safety and tolerability of ZD1839/Nolvadex to placebo/Nolvadex | Safety (frequency and severity of adverse events)
To determine steady-state plasma trough concentrations of tamoxifen in all patients and to compare between the ZD1839/Nolvadex and placebo/Nolvadex treatment arms | Tamoxifen (Cmin) steady-state plasma concentration
To determine steady-state plasma trough concentrations of ZD1839 and relate values to historical data | ZD1839 (Cmin) steady-state plasma concentration
To relate steady-state plasma trough concentrations of ZD1839 to demographic, response, and safety variables | ZD1839 (Cmin) steady-state plasma concentration
To assess the quality of life (QOL) and symptom relief based on the Functional Assessment of Cancer Therapy - Breast (FACT-B) on both treatment arms | FACT-B questionnaire, FBSI (FACT-B Symptom Index)
To investigate subject hospital resource use and health status | Hospitalisations and EQ-5D
Characterization of specific adverse events | Characterization of adverse events such as alopecia, rash and diarrhea
To obtain tumour tissue for biologic studies in this patient population | ER receptor, ErbB-1 &2 (immunohistochemistry) and other biological markers including Her2/neu, AIB1

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Iressa Medical Science Director, MD, Study Director — AstraZeneca
Locations (55):
- United States (4):
  - Research Site, Berkeley, California
  - Research Site, Palm Springs, California
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
- Argentina (9):
  - Research Site, Bahía Blanca
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, El Palomar
  - Research Site, Resistencia
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
  - Research Site, Vicente López
- Australia (5):
  - Research Site, Bentleigh East
  - Research Site, Newcastle
  - Research Site, Randwick
  - Research Site, Westmead
  - Research Site, Wodonga
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Wilrijk
- Brazil (4):
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Saint John, New Brunswick
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Research Site, Herlev, Denmark
- France (4):
  - Research Site, Lyon
  - Research Site, Mougins
  - Research Site, Poitiers
  - Research Site, Rouen
- Germany (5):
  - Research Site, Frankfurt
  - Research Site, Jena
  - Research Site, Kiel
  - Research Site, München
  - Research Site, Trier
- South Africa (4):
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Klerksdorp
  - Research Site, Observatory
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Zaragoza
- United Kingdom (4):
  - Research Site, Colchester
  - Research Site, Dundee
  - Research Site, Manchester
  - Research Site, Nottingham

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1534&filename=CSR-1839IL-0225.pdf